CLINICAL TRIAL: NCT02914613
Title: A Phase I/II Randomized, Double-Masked, Multicenter Clinical Trial Designed to Evaluate the Safety and Exploratory Efficacy of SF0166 Topical Ophthalmic Solution in the Treatment of Diabetic Macular Edema (DME)
Brief Title: Safety and Exploratory Efficacy Study of SF0166 for the Treatment of Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OcuTerra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SF0166-C-001
Record Dates: First submitted 2016-09-01; First posted 2016-09-26 (Estimated); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SF0166 low dose BID (Experimental): SF0166 low dose instilled in study eye BID for 28 days of treatment.
  Interventions: Drug: SF0166 Topical Ophthalmic Solution
- SF0166 high dose BID (Experimental): SF0166 high dose instilled in study eye BID for 28 days of treatment.
  Interventions: Drug: SF0166 Topical Ophthalmic Solution

INTERVENTIONS:
Drug: SF0166 Topical Ophthalmic Solution
  Other Names: OTT166 Ophthalmic Solution

SUMMARY:
The primary purpose of this study was to evaluate the safety and exploratory efficacy of SF0166 Topical Ophthalmic Solution in patients with Diabetic Macular Edema (DME).

DETAILED DESCRIPTION:
This was a prospective, randomized, double-masked, multicenter, Phase I/II clinical study in which 44 eligible subjects with active Diabetic Macular Edema (DME) were randomized to 1 of 2 treatment arms in a 1:1 ratio as follows: SF0166 low dose twice daily (BID) or SF0166 high dose BID.

Study subjects administered the randomly assigned treatment for 28 days. There was an additional 28-day post-treatment follow-up period. Study subjects returned for examination every 2 weeks for 8 weeks (2 months).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older.
2. Retinal thickening secondary to type 1 or type 2 diabetes mellitus with Diabetic Macular Edema (DME) defined as central subfield thickness ≥325 microns (µm) on spectral domain OCT in the study eye.
3. Best-corrected Visual Acuity (BCVA) between 78 and 25 letters, inclusive, in the study eye at the screening/randomization visit using Early Treatment Diabetic Retinopathy Study (ETDRS) testing, with BCVA decrement primarily attributable to Diabetic Macular Edema (DME).
4. Treatment naïve (i.e., no previous anti--vascular endothelial growth factor [VEGF] treatment in the study eye) or previously treated study eye with adequate washout defined below:

   1. Lucentis (ranibizumab): 30-day washout
   2. Avastin (bevacizumab): 30-day washout
   3. Eylea (aflibercept): 60-day washout
   4. Macugen (pegaptanib): 45-day washout
5. Willing and able to return for all study visits.
6. Able to adhere to the study dosing requirements.
7. Understands and signs the written informed consent form.

Exclusion Criteria:

1. Active proliferative diabetic retinopathy (PDR) in the study eye, such as neovascularization of the optic disc (NVD), neovascularization elsewhere (NVE), vitreous hemorrhage, or neovascular glaucoma.
2. Uncontrolled glaucoma or ocular hypertension in the study eye defined as an intraocular pressure (IOP) >25 millimeter of mercury (mmHg) regardless of concomitant treatment with IOP-lowering medications.
3. Uncontrolled hypertension defined as systolic >180 mmHg or >160 mmHg on 2 consecutive measurements (during the same visit) or diastolic >100 mmHg on optimal medical regimen.
4. Screening glycated hemoglobin (HbA1c) blood test >12.0%.
5. Previous panretinal photocoagulation (PRP) in the study eye within 4 months of study enrollment, or the need for PRP during the study based on the Investigator's opinion.
6. Previous focal laser photocoagulation in the study eye, within the foveal avascular zone.
7. Intravitreal/periocular/topical ocular steroids of any type in the study eye within 90 days (3 months) prior to study enrollment.
8. Placement of Iluvien or Retisert (fluocinolone acetonide intravitreal implant) in the study eye within 36 months (3 years) prior to study enrollment.
9. Use of Ozurdex (dexamethasone intravitreal implant) in the study eye within 180 days (6 months) prior to study enrollment.
10. Significant epiretinal membrane, posterior hyaloidal traction, and/or vitreomacular traction in the study eye as determined by the optical coherence tomography (OCT) results.
11. Previous pars plana vitrectomy in the study eye.
12. Any intraocular surgery in the study eye within 90 days (3 months) prior to study enrollment.
13. Yttrium aluminium garnet (YAG) laser treatment in the study eye within 30 days (1 month) prior to study enrollment.
14. Concomitant use of any topical ophthalmic medications in the study eye, including dry eye or glaucoma medications, unless on a stable dose for at least 90 days (3 months) prior to study enrollment and expected to stay on stable dose throughout study participation. Artificial tears are allowed.
15. High myopia in the study eye, with a spherical equivalent of >8.00 Diopters (D) at screening.
16. Chronic or recurrent uveitis in the study eye.
17. Ongoing ocular infection or inflammation in either eye.
18. A history of cataract surgery complicated by vitreous loss in the study eye.
19. Congenital eye malformations in the study eye.
20. A history of penetrating ocular trauma in the study eye.
21. Mentally handicapped.
22. Females of childbearing potential (i.e., who are not postmenopausal for at least 1 year or surgically sterile for at least 6 weeks prior to Visit 1 - Screening/Randomization) who are lactating, or who are pregnant as determined by a positive urine pregnancy test (UPT) at Visit 1 - Screening/Randomization. Women of childbearing potential must agree to use acceptable methods of birth control throughout the study. Acceptable methods of birth control include tubal ligation, transdermal patch, intrauterine devices/systems, oral/implantable/injectable or contraceptives, sexual abstinence, double barrier method, or vasectomized partner.
23. Participation in any other investigational device or drug clinical research study within 30 days of Visit 1 - Screening/Randomization.
24. Contraindication to the study medications or fluorescein dye.
25. Other ocular pathologies that in the Investigator's opinion would interfere with the subject's vision in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foulks, MD, Study Chair — Medical Monitor
Locations (6):
- United States (6):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - United Medical Research Institute, Inglewood, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- SF0166 Low Dose 2.5% BID: SF0166 low dose 2.5% instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
- SF0166 High Dose 5.0% BID: SF0166 high dose 5.0% instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
Period: Overall Study
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Started | 22 | 22
Completed | 20 | 20
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SF0166 High Dose 5% BID: SF0166 high dose 5.0% instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
- Total: Total of all reporting groups
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5% BID | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (13.6) | 67.2 (9.8) | 66.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 11 | 15 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 13 | 19 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Iris Color [Count of Participants; unit: Participants]
  Blue | 4 | 10 | 14
  Brown | 14 | 10 | 24
  Green | 2 | 1 | 3
  Hazel | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With No Cells Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Percentage of subjects with red blood cell counts in the anterior chamber in the ranges from 0 to > 30 with the higher number being worse
Time Frame: Baseline, 2, 4, 6, and 8 weeks
Population: The analysis population at Baseline includes all randomized participants, 22 in each group. Before Week 2, there were two discontinuations, one in each group. Before Week 4 there was one discontinuation in the high dose 5.0% group. One participant in each dose group missed the Week 4 visit. Prior to Week 6 there was one discontinuation in the low dose 2.5% group. One low dose 2.5% group participant missed the Week 6 visit. At Week 8, all the non-discontinued were assessed, 20 in each dose group.
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye) - No cells seen | 22 | 22
  Baseline (Fellow Eye) - No cells seen | 22 | 22
  Week 2 (Study Eye) - No cells seen: number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye) - No cells seen | 21 | 21
  Week 2 (Fellow Eye) - No cells seen: number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye) - No cells seen | 21 | 21
  Week 4 (Study Eye) - No cells seen: number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye) - No cells seen | 20 | 19
  Week 4 (Fellow Eye) - No cells seen: number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye) - No cells seen | 20 | 19
  Week 6 (Study Eye) - No cells seen: number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye) - No cells seen | 19 | 20
  Week 6 (Fellow Eye) - No cells seen: number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye) - No cells seen | 19 | 20
  Week 8 (Study Eye) - No cells seen: number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye) - No cells seen | 20 | 20
  Week 8 (Fellow Eye) - No cells seen: number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye) - No cells seen | 20 | 20

2. Primary Outcome: Number of Subjects With Flare Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with flare in the anterior chamber graded on a scale from 0 (none) to 4 (severe).
Time Frame: Baseline, 2, 4, 6, and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- SF0166 High Dose 5.0% BID: SF0166 high dose 5.0 % instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye) | 0 | 0
  Baseline (Fellow Eye) | 0 | 0
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye) | 0 | 0
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye) | 0 | 0
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye) | 0 | 0
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye) | 0 | 0
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye) | 0 | 0
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye) | 0 | 0
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye) | 0 | 0
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye) | 0 | 0

3. Primary Outcome: Number of Subjects With Hyphema Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with hyphema
Time Frame: Baseline, 2, 4, 6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Mild | 0 | 0
  Baseline (Study Eye): Absent | 22 | 22
  Baseline (Fellow Eye): Mild | 0 | 0
  Baseline (Fellow Eye): Absent | 22 | 22
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Mild | 0 | 0
  Week 2 (Study Eye): Absent | 21 | 21
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Mild | 0 | 0
  Week 2 (Fellow Eye): Absent | 21 | 21
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Mild | 0 | 0
  Week 4 (Study Eye): Absent | 20 | 19
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Mild | 0 | 0
  Week 4 (Fellow Eye): Absent | 20 | 19
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Mild | 0 | 0
  Week 6 (Study Eye): Absent | 19 | 20
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Mild | 1 | 0
  Week 6 (Fellow Eye): Absent | 18 | 20
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Mild | 0 | 0
  Week 8 (Study Eye): Absent | 20 | 20
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Mild | 0 | 0
  Week 8 (Fellow Eye): Absent | 20 | 20

4. Primary Outcome: Number of Subjects With Bulbar Conjunctival Injection Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with bulbar conjunctival injection
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Mild | 0 | 0
  Baseline (Study Eye): Absent | 22 | 22
  Baseline (Fellow Eye): Mild | 0 | 1
  Baseline (Fellow Eye): Absent | 22 | 21
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Mild | 0 | 0
  Week 2 (Study Eye): Absent | 21 | 21
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Mild | 0 | 0
  Week 2 (Fellow Eye): Absent | 21 | 21
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Mild | 0 | 0
  Week 4 (Study Eye): Absent | 20 | 19
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Mild | 0 | 0
  Week 4 (Fellow Eye): Absent | 20 | 19
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Mild | 0 | 0
  Week 6 (Study Eye): Absent | 19 | 20
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Mild | 0 | 0
  Week 6 (Fellow Eye): Absent | 19 | 20
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Mild | 0 | 0
  Week 8 (Study Eye): Absent | 20 | 20
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Mild | 0 | 0
  Week 8 (Fellow Eye): Absent | 20 | 20

5. Primary Outcome: Number of Subjects With Erythema Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with erythema
Time Frame: Baseline, 2, 4, 6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Mild | 0 | 0
  Baseline (Study Eye): Absent | 22 | 22
  Baseline (Fellow Eye): Mild | 0 | 1
  Baseline (Fellow Eye): Absent | 22 | 21
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Mild | 0 | 0
  Week 2 (Study Eye): Absent | 21 | 21
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Mild | 0 | 0
  Week 2 (Fellow Eye): Absent | 21 | 21
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Mild | 0 | 0
  Week 4 (Study Eye): Absent | 20 | 19
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Mild | 0 | 0
  Week 4 (Fellow Eye): Absent | 20 | 19
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Mild | 0 | 0
  Week 6 (Study Eye): Absent | 19 | 20
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Mild | 0 | 0
  Week 6 (Fellow Eye): Absent | 19 | 20
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Mild | 0 | 0
  Week 8 (Study Eye): Absent | 20 | 20
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Mild | 0 | 0
  Week 8 (Fellow Eye): Absent | 20 | 20

6. Primary Outcome: Number of Subjects With Edema Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with edema
Time Frame: Baseline, 2,4, 6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Moderate | 0 | 0
  Baseline (Study Eye): Mild | 1 | 0
  Baseline (Study Eye): Absent | 21 | 22
  Baseline (Fellow Eye): Moderate | 1 | 0
  Baseline (Fellow Eye): Mild | 0 | 1
  Baseline (Fellow Eye): Absent | 21 | 21
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Moderate | 0 | 0
  Week 2 (Study Eye): Mild | 1 | 0
  Week 2 (Study Eye): Absent | 20 | 21
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Moderate | 1 | 0
  Week 2 (Fellow Eye): Mild | 0 | 0
  Week 2 (Fellow Eye): Absent | 20 | 21
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Moderate | 0 | 0
  Week 4 (Study Eye): Mild | 0 | 0
  Week 4 (Study Eye): Absent | 20 | 19
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Moderate | 0 | 0
  Week 4 (Fellow Eye): Mild | 0 | 0
  Week 4 (Fellow Eye): Absent | 20 | 19
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Moderate | 0 | 0
  Week 6 (Study Eye): Mild | 0 | 0
  Week 6 (Study Eye): Absent | 19 | 20
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Moderate | 0 | 0
  Week 6 (Fellow Eye): Mild | 0 | 0
  Week 6 (Fellow Eye): Absent | 19 | 20
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Moderate | 0 | 0
  Week 8 (Study Eye): Mild | 0 | 0
  Week 8 (Study Eye): Absent | 20 | 20
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Moderate | 0 | 0
  Week 8 (Fellow Eye): Mild | 0 | 0
  Week 8 (Fellow Eye): Absent | 20 | 20

7. Primary Outcome: Number of Subjects With Any Lens Opacity Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with any lens opacity
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Any opacity in the lens | 13 | 7
  Baseline (Study Eye): No opacity in the lens | 9 | 15
  Baseline (Fellow Eye): Any opacity in the lens | 15 | 9
  Baseline (Fellow Eye): No opacity in the lens | 7 | 13
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Any opacity in the lens | 12 | 7
  Week 2 (Study Eye): No opacity in the lens | 9 | 14
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Any opacity in the lens | 14 | 8
  Week 2 (Fellow Eye): No opacity in the lens | 7 | 13
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Any opacity in the lens | 13 | 8
  Week 4 (Study Eye): No opacity in the lens | 7 | 11
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Any opacity in the lens | 14 | 8
  Week 4 (Fellow Eye): No opacity in the lens | 6 | 11
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Any opacity in the lens | 10 | 7
  Week 6 (Study Eye): No opacity in the lens | 9 | 13
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Any opacity in the lens | 12 | 7
  Week 6 (Fellow Eye): No opacity in the lens | 7 | 13
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Any opacity in the lens | 11 | 8
  Week 8 (Study Eye): No opacity in the lens | 9 | 12
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Any opacity in the lens | 13 | 7
  Week 8 (Fellow Eye): No opacity in the lens | 7 | 13

8. Primary Outcome: Number of Subjects With Abnormal Findings in Optic Nerve Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the optic nerve
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Normal | 21 | 22
  Baseline (Study Eye): Abnormal | 1 | 0
  Baseline (Fellow Eye): Normal | 20 | 21
  Baseline (Fellow Eye): Abnormal | 2 | 1
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Normal | 21 | 21
  Week 2 (Study Eye): Abnormal | 0 | 0
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Normal | 20 | 20
  Week 2 (Fellow Eye): Abnormal | 1 | 1
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Normal | 20 | 19
  Week 4 (Study Eye): Abnormal | 0 | 0
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Normal | 19 | 19
  Week 4 (Fellow Eye): Abnormal | 1 | 0
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Normal | 19 | 20
  Week 6 (Study Eye): Abnormal | 0 | 0
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Normal | 18 | 20
  Week 6 (Fellow Eye): Abnormal | 1 | 0
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Normal | 20 | 20
  Week 8 (Study Eye): Abnormal | 0 | 0
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Normal | 19 | 20
  Week 8 (Fellow Eye): Abnormal | 1 | 0

9. Primary Outcome: Number of Subjects With Abnormal Findings in Vitreous Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects (both eyes) with abnormal findings in the vitreous
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Normal | 18 | 16
  Baseline (Study Eye): Abnormal | 4 | 6
  Baseline (Fellow Eye): Normal | 17 | 16
  Baseline (Fellow Eye): Abnormal | 5 | 6
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Normal | 16 | 15
  Week 2 (Study Eye): Abnormal | 5 | 6
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Normal | 16 | 16
  Week 2 (Fellow Eye): Abnormal | 5 | 5
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Normal | 16 | 14
  Week 4 (Study Eye): Abnormal | 4 | 5
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Normal | 15 | 14
  Week 4 (Fellow Eye): Abnormal | 5 | 5
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Normal | 15 | 15
  Week 6 (Study Eye): Abnormal | 4 | 5
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Normal | 16 | 15
  Week 6 (Fellow Eye): Abnormal | 3 | 5
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Normal | 17 | 17
  Week 8 (Study Eye): Abnormal | 3 | 3
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Normal | 15 | 16
  Week 8 (Fellow Eye): Abnormal | 5 | 4

10. Primary Outcome: Number of Subjects With Abnormal Findings in Fundus Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the fundus
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Normal | 5 | 8
  Baseline (Study Eye): Abnormal | 17 | 14
  Baseline (Fellow Eye): Normal | 4 | 8
  Baseline (Fellow Eye): Abnormal | 18 | 14
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Normal | 4 | 6
  Week 2 (Study Eye): Abnormal | 17 | 15
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Normal | 4 | 6
  Week 2 (Fellow Eye): Abnormal | 17 | 15
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Normal | 4 | 6
  Week 4 (Study Eye): Abnormal | 16 | 13
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Normal | 4 | 6
  Week 4 (Fellow Eye): Abnormal | 16 | 13
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Normal | 4 | 6
  Week 6 (Study Eye): Abnormal | 15 | 14
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Normal | 4 | 6
  Week 6 (Fellow Eye): Abnormal | 15 | 14
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Normal | 4 | 6
  Week 8 (Study Eye): Abnormal | 16 | 14
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Normal | 4 | 6
  Week 8 (Fellow Eye): Abnormal | 16 | 14

11. Primary Outcome: Number of Subjects With Abnormal Findings in Macula/Choroid Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the macula/choroid
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Abnormal | 22 | 22
  Baseline (Study Eye): Normal | 0 | 0
  Baseline (Fellow Eye): Abnormal | 21 | 22
  Baseline (Fellow Eye): Normal | 1 | 0
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Abnormal | 21 | 21
  Week 2 (Study Eye): Normal | 0 | 0
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Abnormal | 20 | 21
  Week 2 (Fellow Eye): Normal | 1 | 0
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Abnormal | 20 | 19
  Week 4 (Study Eye): Normal | 0 | 0
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Abnormal | 19 | 19
  Week 4 (Fellow Eye): Normal | 1 | 0
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Abnormal | 19 | 20
  Week 6 (Study Eye): Normal | 0 | 0
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Abnormal | 18 | 20
  Week 6 (Fellow Eye): Normal | 1 | 0
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Abnormal | 20 | 20
  Week 8 (Study Eye): Normal | 0 | 0
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Abnormal | 19 | 20
  Week 8 (Fellow Eye): Normal | 1 | 0

12. Primary Outcome: Number of Subjects With Abnormal Findings in Vessels Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the retinal vessels
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Abnormal | 18 | 15
  Baseline (Study Eye): Normal | 4 | 7
  Baseline (Fellow Eye): Abnormal | 17 | 17
  Baseline (Fellow Eye): Normal | 5 | 5
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): Abnormal | 18 | 16
  Week 2 (Study Eye): Normal | 3 | 5
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): Abnormal | 17 | 17
  Week 2 (Fellow Eye): Normal | 4 | 4
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): Abnormal | 17 | 15
  Week 4 (Study Eye): Normal | 3 | 4
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): Abnormal | 16 | 15
  Week 4 (Fellow Eye): Normal | 4 | 4
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): Abnormal | 16 | 16
  Week 6 (Study Eye): Normal | 3 | 4
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): Abnormal | 15 | 16
  Week 6 (Fellow Eye): Normal | 4 | 4
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): Abnormal | 18 | 16
  Week 8 (Fellow Eye): Normal | 2 | 4
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): Abnormal | 18 | 16
  Week 8 (Study Eye): Normal | 2 | 4

13. Primary Outcome: Cup:Disc Ratio of Subjects Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with specified Cup:Disc ratio in the range from 0.1 to 0.6 with the higher number being worse
Time Frame: Baseline, 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): 0.10 | 1 | 4
  Baseline (Study Eye): 0.20 | 6 | 3
  Baseline (Study Eye): 0.30 | 9 | 10
  Baseline (Study Eye): 0.35 | 1 | 0
  Baseline (Study Eye): 0.40 | 2 | 4
  Baseline (Study Eye): 0.50 | 3 | 1
  Baseline (Study Eye): 0.60 | 0 | 0
  Baseline (Fellow Eye): 0.10 | 1 | 3
  Baseline (Fellow Eye): 0.20 | 6 | 3
  Baseline (Fellow Eye): 0.30 | 10 | 13
  Baseline (Fellow Eye): 0.35 | 1 | 0
  Baseline (Fellow Eye): 0.40 | 2 | 3
  Baseline (Fellow Eye): 0.50 | 1 | 0
  Baseline (Fellow Eye): 0.60 | 1 | 0
  Week 2 (Study Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Study Eye): 0.10 | 1 | 4
  Week 2 (Study Eye): 0.20 | 6 | 2
  Week 2 (Study Eye): 0.30 | 8 | 10
  Week 2 (Study Eye): 0.35 | 1 | 0
  Week 2 (Study Eye): 0.40 | 2 | 4
  Week 2 (Study Eye): 0.50 | 3 | 1
  Week 2 (Study Eye): 0.60 | 0 | 0
  Week 2 (Fellow Eye): number analyzed (Participants) | 21 | 21
  Week 2 (Fellow Eye): 0.10 | 1 | 3
  Week 2 (Fellow Eye): 0.20 | 6 | 2
  Week 2 (Fellow Eye): 0.30 | 10 | 13
  Week 2 (Fellow Eye): 0.35 | 1 | 0
  Week 2 (Fellow Eye): 0.40 | 1 | 3
  Week 2 (Fellow Eye): 0.50 | 1 | 0
  Week 2 (Fellow Eye): 0.60 | 1 | 0
  Week 4 (Study Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Study Eye): 0.10 | 1 | 3
  Week 4 (Study Eye): 0.20 | 5 | 1
  Week 4 (Study Eye): 0.30 | 8 | 10
  Week 4 (Study Eye): 0.35 | 1 | 0
  Week 4 (Study Eye): 0.40 | 2 | 4
  Week 4 (Study Eye): 0.50 | 3 | 1
  Week 4 (Study Eye): 0.60 | 0 | 0
  Week 4 (Fellow Eye): number analyzed (Participants) | 20 | 19
  Week 4 (Fellow Eye): 0.10 | 1 | 3
  Week 4 (Fellow Eye): 0.20 | 5 | 1
  Week 4 (Fellow Eye): 0.30 | 10 | 12
  Week 4 (Fellow Eye): 0.35 | 1 | 0
  Week 4 (Fellow Eye): 0.40 | 1 | 3
  Week 4 (Fellow Eye): 0.50 | 1 | 0
  Week 4 (Fellow Eye): 0.60 | 1 | 0
  Week 6 (Study Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Study Eye): 0.10 | 1 | 3
  Week 6 (Study Eye): 0.20 | 6 | 2
  Week 6 (Study Eye): 0.30 | 7 | 10
  Week 6 (Study Eye): 0.35 | 1 | 0
  Week 6 (Study Eye): 0.40 | 1 | 4
  Week 6 (Study Eye): 0.50 | 3 | 1
  Week 6 (Study Eye): 0.60 | 0 | 0
  Week 6 (Fellow Eye): number analyzed (Participants) | 19 | 20
  Week 6 (Fellow Eye): 0.10 | 1 | 3
  Week 6 (Fellow Eye): 0.20 | 6 | 2
  Week 6 (Fellow Eye): 0.30 | 9 | 12
  Week 6 (Fellow Eye): 0.35 | 1 | 0
  Week 6 (Fellow Eye): 0.40 | 0 | 3
  Week 6 (Fellow Eye): 0.50 | 1 | 0
  Week 6 (Fellow Eye): 0.60 | 1 | 0
  Week 8 (Study Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Study Eye): 0.10 | 1 | 3
  Week 8 (Study Eye): 0.20 | 6 | 2
  Week 8 (Study Eye): 0.30 | 7 | 10
  Week 8 (Study Eye): 0.35 | 1 | 0
  Week 8 (Study Eye): 0.40 | 2 | 4
  Week 8 (Study Eye): 0.50 | 3 | 1
  Week 8 (Study Eye): 0.60 | 0 | 0
  Week 8 (Fellow Eye): number analyzed (Participants) | 20 | 20
  Week 8 (Fellow Eye): 0.10 | 1 | 3
  Week 8 (Fellow Eye): 0.20 | 6 | 2
  Week 8 (Fellow Eye): 0.30 | 9 | 12
  Week 8 (Fellow Eye): 0.35 | 1 | 0
  Week 8 (Fellow Eye): 0.40 | 1 | 3
  Week 8 (Fellow Eye): 0.50 | 1 | 0
  Week 8 (Fellow Eye): 0.60 | 1 | 0

14. Primary Outcome: Number of Subjects With Abnormal Findings Following A Fluorescein Angiogram at Week 4 Compared to Baseline (Day 0)
Description: Number and percentage of subjects with abnormal fluorescein angiogram findings
Time Frame: Baseline and 4 weeks
Population: The analysis population at Baseline includes all randomized participants, 22 in each group. The only planned subsequent assessment was at Week 4, end of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
Participants
  Baseline (Study Eye): Abnormal | 21 | 20
  Baseline (Study Eye): Normal | 1 | 2
  Baseline (Fellow Eye): Abnormal | 21 | 19
  Baseline (Fellow Eye): Normal | 1 | 3
  Week 4 (Study Eye): number analyzed (Participants) | 19 | 19
  Week 4 (Study Eye): Abnormal | 18 | 18
  Week 4 (Study Eye): Normal | 1 | 1
  Week 4 (Fellow Eye): number analyzed (Participants) | 19 | 19
  Week 4 (Fellow Eye): Abnormal | 18 | 18
  Week 4 (Fellow Eye): Normal | 1 | 1

15. Primary Outcome: Change in Intraocular Pressure From Baseline to Week 8
Description: Mean and standard deviation of change from Baseline in intra-ocular pressure
Time Frame: 2,4,6 and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 22
mmHg
  Change from Baseline in Study Eye at Week 2: number analyzed (Participants) | 21 | 21
  Change from Baseline in Study Eye at Week 2 | -0.1 (2.5) | 1.0 (3.4)
  Change from Baseline in Non-Study Eye at Week 2: number analyzed (Participants) | 21 | 21
  Change from Baseline in Non-Study Eye at Week 2 | 0.2 (2.6) | -0.1 (2.8)
  Change from Baseline in Study Eye at Week 4: number analyzed (Participants) | 20 | 19
  Change from Baseline in Study Eye at Week 4 | -0.2 (3.1) | 1.2 (2.4)
  Change from Baseline in Non-Study Eye at Week 4: number analyzed (Participants) | 20 | 19
  Change from Baseline in Non-Study Eye at Week 4 | 0.2 (3.1) | 0.3 (2.6)
  Change from Baseline in Study Eye at Week 6: number analyzed (Participants) | 19 | 20
  Change from Baseline in Study Eye at Week 6 | -0.3 (2.9) | 0.2 (2.5)
  Change from Baseline in Non-Study Eye at Week 6: number analyzed (Participants) | 19 | 20
  Change from Baseline in Non-Study Eye at Week 6 | 0.3 (2.3) | -0.5 (3.2)
  Change from Baseline in Study Eye at Week 8: number analyzed (Participants) | 20 | 20
  Change from Baseline in Study Eye at Week 8 | -0.2 (2.8) | 1.0 (2.0)
  Change from Baseline in Non-Study Eye at Week 8: number analyzed (Participants) | 20 | 20
  Change from Baseline in Non-Study Eye at Week 8 | 0.6 (3.2) | -0.9 (2.7)

16. Primary Outcome: Change in Central Retinal Thickness (CRT) for Study Eye From Baseline (Day 0) to Week 8
Time Frame: 2,4,6 and 8 weeks
Population: The analysis population is the per protocol population with 19 participants in each dose group at Baseline. One participant in each group missed the Week 4 visit and one participant in the low dose 2.5% group missed the Week 6 visit. Four participants, three in the low dose group and one in the high dose group, were administered rescue medication at clinic visits and their data from subsequent visits are excluded. One participant in each dose group was excluded for having an out-of-window visit.
Measure: Mean (Standard Deviation); unit: change from baseline
Groups:
- SF0166 Low Dose 2.5% BID: SF0166 low dose 2.5% will be instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
- SF0166 High Dose 5.0% BID: SF0166 high dose 5.0% will be instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 19 | 19
change from baseline
  Change from Baseline at Week 2 | 24.9 (117.3) | 1.3 (56.5)
  Change from Baseline at Week 4: number analyzed (Participants) | 18 | 18
  Change from Baseline at Week 4 | 17.0 (125.6) | 3.4 (49.5)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 19
  Change from Baseline at Week 6 | -16.3 (71.1) | 14.9 (84.5)
  Change from Baseline at Week 8: number analyzed (Participants) | 15 | 17
  Change from Baseline at Week 8 | -46.5 (101.2) | 14.6 (110.3)

17. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) for Study Eye From Baseline (Day 0) at Week 4 and Week 8
Time Frame: 2, 4, 6 and 8 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: change from baseline
Groups:
- SF0166 High Dose 5% BID: SF0166 high dose 5.0% will be instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5% BID
Number analyzed (Participants) | 19 | 19
change from baseline
  Change from Baseline at Week 2 | 0.1 (5.4) | -0.8 (4.3)
  Change from Baseline at Week 4: number analyzed (Participants) | 18 | 18
  Change from Baseline at Week 4 | 0.1 (5.7) | 0.8 (3.5)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 19
  Change from Baseline at Week 6 | 1.1 (6.1) | -0.5 (3.2)
  Change from Baseline at Week 8: number analyzed (Participants) | 15 | 17
  Change from Baseline at Week 8 | 1.6 (5.2) | -0.2 (5.7)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 5/22 | 1/22
Other Adverse Events (participants affected / at risk) | 10/22 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SF0166 Low Dose 2.5% BID (N=22) | SF0166 High Dose 5.0% BID (N=22)
Cardiomyopathy (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SF0166 Low Dose 2.5% BID (N=22) | SF0166 High Dose 5.0% BID (N=22)
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 2
Cataract (Eye disorders) | 0 | 2
Ocular hyperaemia (Eye disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Unevaluable event (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Infections and infestations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT02914613/Prot_SAP_000.pdf